CLINICAL TRIAL: NCT02960568
Title: Genetic Variability in the Cytochrome P-450 Isoenzyme 2D6 (CYP2D6) in an Active Duty U.S. Military Population and the Impact of CYP2D6 Phenotype on Primaquine Metabolism.
Brief Title: Genetic Variability in CYP2D6 in U.S Active Duty Population
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: WR2253; D6.7_14_I_14_J9_837 (Other Grant/Funding Number: Defense Health Program)
Record Dates: First submitted 2016-11-02; First posted 2016-11-09 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Pharmacologic Action
Keywords: primaquine; metabolism; malaria; hypnozoite; vivax; CYP2D6; active duty personnel
MeSH Terms: conditions — Malaria | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primaquine (Experimental): Poor and Intermediate Metabolizers will receive 30 mg oral primaquine (PQ) and have peripheral blood draws over a 24-hour period to measure PQ pharmacokinetics
  Interventions: Drug: Primaquine
- No primaquine (No Intervention): Extensive and Ultra Metabolizers will not be eligible for the pharmacokinetic portion of the study and participation will be complete after receiving genotype information

INTERVENTIONS:
Drug: Primaquine — 30 mg oral primaquine one time
  Arms: Primaquine

SUMMARY:
The investigator proposes to 2D6 (Cytochrome P-450 Isoenzyme 2D6) genotype and phenotype a group of active duty service members and assess the effects on primaquine metabolism.

DETAILED DESCRIPTION:
The investigator propose to enroll a group of active duty service members in order to determine individuals' 2D6 isoenzyme genotype, an enzyme belonging to the hepatic cytochrome P450 oxidase system. The 2D6 isoenzyme is a key enzyme involved in the metabolism of many drugs including the anti-malarial drug primaquine (PQ). By knowing the genotype, the investigator can then categorize each volunteer by CYP2D6 phenotype i.e., expected impact on drug metabolism. In order to further substantiate the relationship between CYP2D6 activity, inadequate metabolism and subsequent primaquine failure, the investigator proposes to assess the effect of 2D6 genetic polymorphisms on PQ metabolism by measuring the PQ pharmacokinetics (PK) over 24 hours following a single 30 mg oral dose in a subset of these Active Duty subjects.

ELIGIBILITY:
Inclusion criteria:

* Active duty Service member, (male or female) 18 to 60 years of age (inclusive) at the time of enrollment
* Written informed consent for phase 1 must be obtained
* Written informed consent for phase 2 must be obtained from the subject before the screening procedures
* Free of significant health problems as established by medical history, laboratory and clinical examination before entering the study
* If the subject is female, she must be of non-childbearing potential (either surgically sterilized or one year post-menopausal) or, if of childbearing potential, she must be capable of preventing pregnancy, have a negative pregnancy test at the time of the administration of primaquine , and must agree to continue such precautions until 48 hours after primaquine administration.
* Normal (non-deficient) G6PD (glucose-6-phosphate dehydrogenase) phenotype (range: 4.6 to 13.5 units/gm hemoglobin)
* Subjects must obtain approval from his or her supervisor per Walter Reed Army Institute of Research (WRAIR) Policy 06-15 in order to be participate in the PQ PK portion of phase 2

Exclusion criteria:

* Use of any investigational or non-registered drug within 30 days preceding the primaquine dosing.
* Pregnant (positive urine β-HCG) or nursing at screening or plans to become pregnant or nurse from the time of enrollment until 48 hours after primaquine dosing.
* Allergy to primaquine
* Use of medications known to cause drug interactions with primaquine or CYP2D6
* Acute or chronic, clinically significant, pulmonary, cardiovascular, hepatic, neurologic, or renal functional abnormality, as determined by history, physical examination, and laboratory evaluation
* History of hemolytic anemia
* Any abnormal baseline laboratory screening tests listed below (normal values are defined by the current Quest Diagnostics reference guide on file in the CTC):

  * ALT (alanine aminotransferase)above normal range
  * Glomerular filtration rate (GFR) below normal range for the subject's ethnicity
  * Hemoglobin below normal range
* Hepatomegaly, right upper quadrant abdominal pain or tenderness
* Suspected or known current alcohol abuse as determined from the medical history or by physical examination
* Use of any drugs that may cause hemolytic anemia and/or bone marrow suppression such as quinacrine, dapsone, rifampin, colchicine, ribavirin, penicillamine and sulfonamides.
* Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 550 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Description of CYP2D6 alleles in an active duty population | 1 hour
  Genotyping of CYP2D6 alleles will be analyzed by a multiplexed cytometric bead array assay, Luminex xTAG® CYP2D6 Kit v3 (Austin, TX) which allows for detection of the 16 major alleles of 2D6 in the United States: 1,2,3,4,5,6,7,8,9,10,11,15, 17,29, 35,41. Subjects will then be categorized by CYP2D6 phenotype according to standard definitions of enzyme metabolic activity of specific 2D6 alleles using the published activity score model: AS Model A (1): "poor" (PM), "intermediate" (IM), "extensive" (EM) or "ultra (UM)" enzyme activity compared to the general population. Alleles known to have no activity are scored "0", intermediate activity alleles are scored as 0.5, while alleles with normal activity are scored as 1. Scores of both alleles making up the genotype are then added together to give the AS-Model A score and range from 0 to 2, with 0 indicating little or no CYP2D6 activity and 1 or 2 indicating normal levels of CYP2D6. Data will be descriptively analyzed.
Measure concentrations of plasma primaquine and its major metabolites. | 24 hours
Develop pharmacokinetic curves of primaquine and its major metabolites with determinations of Area under the curve (AUC) | 1 month

OTHER OUTCOMES:
Develop pharmacokinetic curves of primaquine and its major metabolites with determinations of maximum concentration (Cmax) | 1 month
Develop pharmacokinetic curves of primaquine and its major metabolites with determinations of time to reach maximum concentration (Tmax) | 1 month
Develop pharmacokinetic curves of primaquine and its major metabolites with determinations of rate constant (kelim) | 1 month
Develop pharmacokinetic curves of primaquine and its major metabolites with determinations of elimination half-life (t1/2), | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Norman Waters, PhD, Study Director — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- WRAIR, Silver Spring, Maryland, United States

REFERENCES:
- [Derived] Spring MD, Sousa JC, Li Q, Darko CA, Morrison MN, Marcsisin SR, Mills KT, Potter BM, Paolino KM, Twomey PS, Moon JE, Tosh DM, Cicatelli SB, Froude JW, Pybus BS, Oliver TG, McCarthy WF, Waters NC, Smith PL, Reichard GA, Bennett JW. Determination of Cytochrome P450 Isoenzyme 2D6 (CYP2D6) Genotypes and Pharmacogenomic Impact on Primaquine Metabolism in an Active-Duty US Military Population. J Infect Dis. 2019 Oct 22;220(11):1761-1770. doi: 10.1093/infdis/jiz386. PMID 31549155